CLINICAL TRIAL: NCT05143476
Title: Serum-Protein-Based Indices for the Progression of Fracture Healing and Nonunion
Acronym: UNION
Status: Active, not recruiting | Type: Observational
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: W81XWH-19-1-0796
Record Dates: First submitted 2021-11-10; First posted 2021-12-03 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Humerus Fractures
Keywords: Limb Fractures; Failure to Progress; Nonunion; Serum Markers
MeSH Terms: conditions — Humeral Fractures; Dystocia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Each 50mL specimen will be divided into 40 mL of whole blood which will be fixed for storage and 10 mL which will be collected for plasma processing. Plasma samples will be used for analysis of up to ~2000 proteins found in plasma circulation in the blood during the learning phase (Aim1). During the validation phase (Aim2) a more restricted target group of 170 proteins will be assayed. The networks of interaction among various multiple inflammatory mediators, systemic response factors to trauma and locally produced proteins at the repair site during callus formation that spill into the serum will be analyzed. Whole blood as fixed for long term storage will be processed per study operating procedures, for future research endeavors directed at total blood immune cell profiling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational group: Follow-up visits will be conducted at 4-6, 7-9, 12-16 and 26-32 weeks, from time of fracture. A participant's doctor will perform routine examination of fracture healing. The assessment will include evaluation of gross fracture site motion and presence or absence of radiographic healing, including a mRUST score.

SUMMARY:
To define a serum protein-based diagnostic for the progression and failure of fracture healing, through the identification of a set of serum proteins that appear at early times of biological healing and show a specific correlation with later radiological and functional signs used to define delayed healing and non-union.

DETAILED DESCRIPTION:
Aim 1 Learning Set: At the earliest time in the study when 10 non-unions have been identified, we will select 10 control patients matched for comorbidities (including a body mass index>40, smoking history, and diabetes) from the group that has been enrolled for comparison to the 10 non-union patients. The proteins showing the most substantial changes in response to either their initial or end point measurements in both healer and non-healer sets will be identified. Temporal clustering and biological assessment tools will be used to identify the biological processes and time frames showing altered serum levels for these markers. A selection process will then use a set of pair wise iterative processes to identify both single markers and multiple marker subsets that show the best correlations to both mRUST and union/nonunion diagnosis prior to the current time that the diagnosis for failed healing is made.

Aim2 Validation Set: As soon as the next group 10 non-union patients are identified a new group of 10 healers will be selected and the target group of protein identified in phase one will be tested for robustness in a second study with this new set of non-healers healers. Assessments of the robustness will be based on level of detection (LOD) and reproducibility of LOD and diagnostic performance. A third assessment will be carried out with the total group of 20 non healers identified in both the first and second phases of the project by rescreening this group against profiles of a final and novel set of 40 new healers. This new set of healers will be selected from the total patient sets of profiles that have been collected across the entire study period and again will be randomly selected and matched for comorbidities. During each subsequent screen we will refine the marker set further taking into account both performance features, qualitative factors related to a protein's biological functions and relationships to the processes of healing, and their correlation to the clinical parameters that we are using to assess progression of healing (union). The last stage of assessment provides an independent technical biochemical/immunological validation for the ten best performing proteins. This assessment will be made using a conventional Western blot assay across a randomized set of 20 profiles from both healers and non-healers who had been previously screened using the microarray format. This last assay is a quality control step for protein identification specification.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature, ages 18-70 (inclusive)
2. Diagnosis of isolated closed extra-articular fractures of the humeral shaft deemed appropriate for closed treatment by immobilization and a sling by the treating physician
3. Approached for consent within two weeks of injury
4. Available for follow up at this treatment facility for at least six months

Exclusion Criteria:

1. Humeral shaft fractures that extend into the articular surface.
2. Pathologic fractures.
3. Additional long bone injuries or fractures of upper or lower extremity that would compromise outcome assessments of single fracture protein levels.
4. Previous retained hardware in humerus from other injuries.
5. Soft tissue injury compromising selected treatment method.
6. Any injury that involved a trauma activation with entry of more than two AIS codes.
7. Fractures with vascular injury.
8. Pregnant women, potentially pregnant, or lactating women
9. Immunocompromised based on the medical record and patient reported use of pharmacological medications that would lead to immunocompromise. (i.e., Anti-TNF therapies, or associated therapies for treatment of various rheumatological conditions.)
10. Unable to comply with postoperative rehabilitation protocols or instructions (i.e., head injury or cognitively impaired).
11. Known metabolic bone disease.
12. Severe problems with maintaining follow-up (e.g., patients who are prisoners or homeless at the time of injury or who are intellectually challenged without adequate family support).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will consent and enroll up to 180 patients who meet the enrollment inclusion exclusion criteria for this study. In this group we anticipate based on our prior clinical data that about 20 patients would experience failed healing (nonunion) providing us with the ability to identify those protein in the serum that are diagnostic for failed healing. Patient enrollment will take place continuously over a three year period with the two stages of the project initiated when the enrollment numbers are met to carry out each aim of the project. When a patient presents with a humerus fracture he or she will be evaluated (according to standard of care) for possible enrollment in the study. The inclusion /exclusion criteria will be reviewed by the treating surgeon.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
Fracture Healing Outcomes and Functional Healing Outcomes | 7-9 week visit
  The primary outcome for the assessment of fracture healing will be assessed by gross motion and mRUST (modified radiograph union score) score greater than or equal to 6. mRUST score ranges from 4-16 where score greater than or equal to 6 is considered as the predictors of progression to union.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Gerstenfeld, PhD, Principal Investigator — Boston University; Renan C Castillo, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No